CLINICAL TRIAL: NCT00305760
Title: A Safety and Efficacy Trial of Lethally Irradiated Allogeneic Pancreatic Tumor Cells Transfected With the GM-CSF Gene in Combination With Erbitux (Cetuximab) for the Treatment of Advanced Pancreatic Adenocarcinoma
Brief Title: Vaccine Therapy, Cyclophosphamide, and Cetuximab in Treating Patients With Metastatic or Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0501; P30CA006973 (NIH); BMS-CA225247
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; duct cell adenocarcinoma of the pancreas; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide, Pancreatic Tumor Vaccine, Cetuximab (Experimental)
  Interventions: Drug: Cetuximab; Biological: Pancreatic tumor vaccine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered at an initial dose of 400 mg/m2, followed by weekly doses of 250 mg/m2 for a total of 6 cycles that last 3 weeks each.
  Other Names: Erbitux
Biological: Pancreatic tumor vaccine — Vaccine will be administered one day after cyclophosphamide (day 1) every three weeks for 6 cycles.
  Other Names: PANC 10.05 pcDNA-1/GM-Neo and PANC 6.03 pcDNA-1/GM-Neo vaccine; GVAX
Drug: Cyclophosphamide — Cyclophosphamide 250 mg/m2 will be administered one day prior to vaccination (day 0) every three weeks for 6 cycles.
  Other Names: Cytoxan

SUMMARY:
RATIONALE: Vaccines made from gene-modified tumor cells may help the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vaccine therapy together with cyclophosphamide and cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works when given together with cyclophosphamide and cetuximab in treating patients with metastatic or locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of pancreatic tumor vaccine, cyclophosphamide, and cetuximab in patients with metastatic or locally advanced adenocarcinoma of the pancreas.

Secondary

* Determine the overall, progression-free, and event-free survival of patients treated with this regimen.
* Correlate specific in vivo parameters of immune response (e.g., mesothelin, prostate stem cell antigen [PSCA], mutated k-ras-specific T-cell responses) with clinical response in patients treated with this regimen.
* Correlate downstream targets of epidermal growth factor receptor (EGFR) signaling (e.g., intratumor expression of Akt, Stat 3 and 5, mesothelin, mutated k-ras, and PSCA) with inhibition by cetuximab in patients treated with this regimen.
* Correlate inhibition of EGFR signaling (e.g., Stat 3 and 5) with improved specific mesothelin, PSCA, and mutated k-ras-specific T-cell responses in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive cyclophosphamide IV on day 0, sargramostim plasmid DNA pancreatic tumor vaccine intradermally on day 1, and cetuximab IV over 1-2 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection and tumor biopsies periodically during study for biomarker correlative studies.

At the completion of study treatment, patients are followed at 3 weeks and then every 4 weeks for 16 weeks.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal adenocarcinoma of the pancreas

  * Mixed adenocarcinoma tumors eligible provided the predominant invasive component of the tumor is adenocarcinoma
* The following histologic diagnoses are not eligible:

  * Adenosquamous
  * Squamous cell
  * Colloid
  * Islet cell
  * Serous or mucinous cystadenoma or cystadenocarcinoma
  * Carcinoid
  * Small or large cell carcinoma
  * Intraductal oncocytic papillary neoplasms
  * Osteoclast-like giant cell tumors
  * Acinar cell carcinoma
  * Pancreatoblastoma
  * Solid pseudopapillary tumors
  * Undifferentiated small cell carcinoma
  * Nonepithelial tumors (sarcoma, gastrointestinal stromal tumor, lymphoma)
  * Adenocarcinomas of the ampulla, distal bile duct, or duodenum
* Metastatic or locally advanced disease that is refractory to standard therapy OR for which patient refused standard therapy
* Measurable disease defined as ≥ 1 lesion unidimensionally measured as ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

  * No nonmeasurable disease only including, but not limited to, the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No known active or untreated brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 90,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2 mg/dL
* ALT and AST ≤ 5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* No active infection
* No uncontrolled medical condition that would potentially increase the risk of toxicities or complications of study therapy
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No active peptic ulcer disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study treatment
* No other malignancy within the past 5 years except for nonmelanomatous skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* HIV negative
* No active autoimmune disease or prior autoimmune disease requiring medical treatment with systemic immunosuppressants including any of the following:

  * Inflammatory bowel disease
  * Systemic vasculitis
  * Scleroderma
  * Psoriasis
  * Multiple sclerosis
  * Hemolytic anemia or immune thrombocytopenia
  * Rheumatoid arthritis
  * Systemic lupus erythematosus
  * Sjögren's syndrome
  * Sarcoidosis
  * Asthma or chronic obstructive pulmonary disease that does not require systemic corticosteroids or routine use of inhaled steroids allowed
* No known or suspected hypersensitivity to sargramostim (GM-CSF), cyclophosphamide, pentastarch, corn, or DMSO
* No prior severe infusion reaction (> grade 3) to a monoclonal antibody

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 1 month since prior adjuvant chemotherapy
* More than 4 weeks since prior surgery except for minor procedures (e.g., dental work, skin biopsy) and biliary stent placement
* No prior surgical procedures affecting absorption
* More than 4 weeks since prior radiotherapy
* More than 1 month since prior participation in an investigational new drug study
* No unresolved chronic toxicity (except alopecia) from prior anticancer therapy
* More than 28 days since prior systemic steroids
* No concurrent systemic steroids or immunosuppressive drugs

  * Topical, inhaled, and intra-articular steroids allowed
* No other concurrent anticancer vaccine therapy
* No other concurrent chemotherapy, immunotherapy, radiotherapy, gene therapy, biologic therapy, or investigational therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Cyclophosphamide, Pancreatic Tumor Vaccine, Cetuximab
Started | 60
Completed | 13
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Safety of Combining the Pancreatic Tumor Vaccine in Sequence With Cyclophosphamide and Erbitux. Safety is Defined as the Number of Treatment-related Grade 3 or 4 Adverse Events Observed in Greater Than 5% of the Patient Population
Time Frame: 7 months
Measure: Number; unit: Adverse Events
Arm/Group | Cyclophosphamide, Pancreatic Tumor Vaccine, Cetuximab
Number analyzed (Participants) | 60
Adverse Events | 2

ADVERSE EVENTS:
Arm/Group | Cyclophosphamide, Pancreatic Tumor Vaccine, Cetuximab
Serious Adverse Events (participants affected / at risk) | 12/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Pancreatic Tumor Vaccine, Cetuximab (N=60)
Infusion reaction, erbitux (General disorders) | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Pancreatic Tumor Vaccine, Cetuximab (N=60)
Lymphopenia (Blood and lymphatic system disorders) | 5
Hypotension (Cardiac disorders) | 3
Arthragia (Musculoskeletal and connective tissue disorders) | 6
Chills (General disorders) | 6
Fatigue (General disorders) | 9
Fever (General disorders) | 17
Flu like symptoms (General disorders) | 10
Blisters (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema, vaccine site (Skin and subcutaneous tissue disorders) | 56
Induration, vaccine site (Skin and subcutaneous tissue disorders) | 58
Pruritis, vaccine site (Skin and subcutaneous tissue disorders) | 47
Tenderness, vaccine site (Skin and subcutaneous tissue disorders) | 49
Pruritis, generalized (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 35
Diarrhea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 12
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes